CLINICAL TRIAL: NCT02935543
Title: Phase 2 Study of CD19-directed Chimeric Antigen Receptor-modified T Cells (CART19) for Adult Patients With Minimal Residual Disease During Upfront Treatment for Acute Lymphoblastic Leukemia
Brief Title: CART19 in Adult Patients With Minimal Residual Disease During Upfront Treatment for ALL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is terminated because of administrative reasons.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC39416, 825668
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2020-01

CONDITIONS: Leukemia, Acute Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CART19 (Experimental): CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRz:41BB administered by IV infusion.
  Interventions: Biological: CART 19

INTERVENTIONS:
Biological: CART 19 — CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRz:41BB administered by IV infusion. Subjects will receive 1-5 x 10^8 transduced CAR T cells as a split dose over three days as follows:Day 1, 10% fraction: 1-5x10^7 CART19 cells, Day 2, 30% fraction: 3x10^7-1.5x10^8 CART19 cells, Day 3, 60% fraction: 6x10^7-3x10^8 CART19 cells

SUMMARY:
This is a single center, single arm, open-label phase 2 study to determine the efficacy of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART19" cells) in adults with minimal residual disease (MRD) during upfront treatment for CD19+ acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19+, B cell Acute Lymphoblastic Leukemia (B-ALL) who have 0.01%≤MRD<10% during upfront treatment
2. Patients must be within 18 months of initial ALL diagnosis
3. Age ≥18 years
4. Adequate organ function defined as:

   1. Creatinine ≤ grade 2
   2. ALT/AST ≤3x upper limit of normal range for age
   3. Direct bilirubin ≤2.0 mg/dl
   4. Adequate pulmonary function defined as ≤ grade 2 dyspnea and ≤ grade 2 hypoxia
   5. Cardiac Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
5. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy.
6. Expression of CD19 on leukemic blasts demonstrated by flow cytometry or immunohistochemistry of bone marrow or peripheral blood
7. Adequate performance status defined as ECOG Performance Status 0 or 1
8. Provides written informed consent
9. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol

Exclusion Criteria:

1. Active, uncontrolled infection
2. Active hepatitis B or hepatitis C
3. HIV Infection
4. Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 2)
5. Subjects with clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of enrollment.
6. Pregnant or nursing (lactating) women
7. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to leukemia or previous leukemia treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CART19
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CART19
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Conversion of Minimal Residual Disease (MRD) to <0.01%
Description: The incidence of conversion of minimal residual disease (MRD) to <0.01% after CART19 therapy in patients with MRD+ ALL during upfront treatment
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | CART19
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Best Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the date of the first CART19 infusion to the date of death due to any reason.
Time Frame: one year
Population: data were not collected
Arm/Group | CART19
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Remission (DOR)
Description: Duration of remission (DOR) is defined as the duration from the date when the response criteria of CR or CRi is first met to the date of relapse or death due to ALL.
Time Frame: one year
Population: data were not collected
Arm/Group | CART19
Number analyzed (Participants) | 0

4. Secondary Outcome: Relapse Free Survival (RFS)
Description: Relapse free survival (RFS) is defined as the duration between the date when the response criteria of CR or CRi is first met to the date of relapse or death due to any cause.
Time Frame: one year
Population: data were not collected
Arm/Group | CART19
Number analyzed (Participants) | 0

5. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival (EFS) is defined as the time from start of the first CART19 infusion to the earliest of the following:
  Death from any cause Relapse
  Treatment failure: Defined as no response in the study and discontinuation from the study due to any of the following reasons:
  * Adverse event(s)
  * Abnormal laboratory value(s)
  * Abnormal test procedure results
  * New cancer therapy (excluding HSCT when performed in CR or CRi)
Time Frame: one year
Population: data were not collected
Arm/Group | CART19
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Manufacturing Products That do Not Meet Release Criteria for Vector Transduction Efficiency, T Cell Product Purity, Viability, Sterility or Due to Tumor Contamination.
Description: Percentage of manufacturing products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, sterility or due to tumor contamination.
Time Frame: prior to day 1
Measure: Number; unit: percentage of products
Arm/Group | CART19
Number analyzed (Participants) | 1
percentage of products | 0

7. Secondary Outcome: Safety and Tolerability of CART19: Frequency and Severity of Adverse Events, Including, But Not Limited to, Cytokine Release Syndrome (CRS) and Macrophage Activation Syndrome (MAS).
Description: Frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS) and macrophage activation syndrome (MAS).
Time Frame: one year
Measure: Number; unit: percentage of participants
Arm/Group | CART19
Number analyzed (Participants) | 1
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CART19
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CART19 (N=1)
gastric necrosis (Gastrointestinal disorders) | 1 (1)
parathesias (Nervous system disorders) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02935543/Prot_SAP_000.pdf